CLINICAL TRIAL: NCT05246930
Title: The Study of Impulse Oscillometry in Inducible Laryngeal Obstruction
Brief Title: Evaluating the Use of a Device Called Impulse Oscillometry in Participants With Vocal Cord Disorders or Asthma
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Steve Nicholas Georas, Professor, University of Rochester
Other Study IDs: STUDY00006861
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Breathing, Mouth; Lung Function Decreased; Vocal Cord Dysfunction; Laryngeal Obstruction; Asthma
MeSH Terms: conditions — Mouth Breathing; Respiratory Insufficiency; Vocal Cord Dysfunction; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Subjects with a diagnosis of vocal cord dysfunction: Subjects with a confirmed or suspected diagnosis of vocal cord dysfunction (also called inducible laryngeal obstruction). Some subjects will have concomitant diagnosis of asthma.
  Interventions: Device: Impulse Oscillometer
- Subjects with diagnosis of asthma: Subjects with physician-diagnosed asthma. Some subjects will have concomitant diagnosis of vocal cord dysfunction.
  Interventions: Device: Impulse Oscillometer

INTERVENTIONS:
Device: Impulse Oscillometer — The tremoFlo C-100 Airwave Oscillometry System is intended to measure respiratory system impedance using the Forced Oscillation Technique (FOT).
  Other Names: THORASYS tremoFlo C-100 Airwave Oscillometry System

SUMMARY:
This study will determine if airway resistance to airflow and pressure, measured by Impulse Oscillometry, is impacted in subjects with vocal cord disorders and whether these measurements are different when compared to subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Vaccinated against COVID-19 or testing negative for COVID-19 by viral PCT within 5 days before testing
* Willingness to perform breathing test
* Must be able to speak and understand English
* Documented diagnosis of asthma, documented clinical diagnosis of vocal cord dysfunction, or undergoing evaluation for vocal cord dysfunction

Exclusion Criteria:

* Unable to provide consent or perform oscillometry test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to one hundred (100) human subjects will be recruited from the following University of Rochester locations: Mary Parkes Center for Asthma, Allergy, and Pulmonary Care, the Pulmonary Clinic at Strong Memorial Hospital, and The Voice Center, an Otolaryngology Clinic at Clinton Woods.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Mean respiratory system impedance | Single measurement, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Parkes Asthma and Allergy Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Donohue P, Connolly M, D'Alfonso M, Jackson G, Grasso LC, Cai X, O'Connell Ferster AP, Schneider GT, Khurana S, Georas SN. Peripheral airways dysfunction measured by oscillometry differentiates asthma from inducible laryngeal obstruction. Respir Med. 2025 Jan;236:107905. doi: 10.1016/j.rmed.2024.107905. Epub 2024 Dec 3. PMID 39631550